CLINICAL TRIAL: NCT05914350
Title: Comparison Between Ultrasound Guided Ozone, Platelet-Rich Plasma or Steroid Injection in the Treatment of Sacroiliitis; a Randomized Double Blinded Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelnaby Ibrahim, Ahmed elmaghrapy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 36264MD46/3/23
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: the Efficacy of Ultrasound Guided Sacroiliac Injection of Ozone, Platelet Rich Plasma (PRP) or Steroid for Treatment of Sacroiliitis
MeSH Terms: interventions — Steroids; Methylprednisolone Acetate; Lidocaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): 40 mg methylprednisolone acetate and 1 mL lidocaine will be injected in sacroiliac joint in first week by ultrasound. While the second and third injections in the second and third weeks will be done by sham injection
  Interventions: Procedure: ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis; Drug: methylprednisolone acetate and lidocaine
- Group 2 (Experimental): 3 mL PRP and 1 mL lidocaine will be injected in sacroiliac joint by ultrasound once/week for 3 weeks
  Interventions: Procedure: ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis; Drug: PRP and lidocaine
- Group 3 (Experimental): 10 ml of medical ozone of 20 μg/ml will be injected in sacroiliac joint by ultrasound once/week for 3 weeks
  Interventions: Procedure: ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis; Drug: medical ozone

INTERVENTIONS:
Procedure: ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis — ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis
Drug: methylprednisolone acetate and lidocaine — 40 mg methylprednisolone acetate and 1 mL lidocaine
  Arms: Group 1
Drug: PRP and lidocaine — 3 mL PRP and 1 mL lidocaine
  Arms: Group 2
Drug: medical ozone — 10 ml of medical ozone
  Arms: Group 3

SUMMARY:
Comparison between ultrasound guided Ozone, platelet-rich plasma or steroid injection in the treatment of sacroiliitis; a Randomized Double Blinded Controlled Study

DETAILED DESCRIPTION:
The sacroiliac joints (SIJ) are the largest axial joints in the human body. By aging, osteoarthritic degeneration occurs to SIJ. SIJ dysfunction typically results from abnormal motion and malalignment of the joint (1).

SIJ pain is one of the differential diagnoses of low back pain. Approximately, 10-25% of these patients will have SIJ dysfunction which should be considered clinically (1, 2). This pain affects physical, psychological and social aspects of the person reducing the work performance. It imposes a huge burden on nations globally (3, 4).

SIJ pain can be a difficult condition to treat and a multidisciplinary approach to treatment including multimodal medical, psychological, physical, and interventional approach is recommended (5).

Corticosteroids are a very magic therapy since their first use and they offer anti-inflammatory mechanisms to reduce low back pain and joint pain. SIJ steroid injections are typically performed for SIJ pain related to osteoarthritis, ligamentous sprain and sacroiliitis associated with inflammatory spondyloarthropathies (5, 6).

Intra-articular steroid injections have intermediate-term benefits, in which more than half of the patients had positive responses to treatment in a 6-month follow-up (7, 8).

Another treatment modality is Platelet-rich plasma (PRP) which is autologous blood that contains platelet concentrations above normal physiological levels (9). PRP is believed to stimulate regeneration through the release of growth factors and proteins that may be involved in repairing the degeneration (10, 11).

While corticostroid injection has rapid onset of pain releif with short duration, the PRP injection has delayed onset and long term of pain releif in recent studies (12-14).

Ozone therapy has been used in the treatment of many musculoskeletal diseases including low back pain (LBP), lumbar disk herniation, cervical pain, cervical disk herniation, failed back surgery syndrome, degenerative spinal disease, knee osteoarthritis, meniscal injuries, sacroiliitis, plantar fasciitis and carpal tunnel syndrome (8, 15). However, ozone therapy is not tested well in SIJ. Ozone has multiple mechanisms of action:, antioxidant, analgesic and antiinflammatory effects (16, 17).

Ultrasound has gained increasing popularity in pain management (18). Furthermore, it is a valuable tool for pain physicians in confirming the diagnosis of many musculoskeletal pain conditions (19). It has many advantages when compared to fluoroscopy techniques (20). It has no radiation exposure, procedures can be done outside operating room which will decrease the costs (21).

ELIGIBILITY:
Inclusion Criteria:

- One hundred and five patients, ASA physical status I - III, age 21 - 65 years, diagnosed with sacroiliitis.

Exclusion Criteria:

* • Patient refusal

  * Psychological disturbance.
  * Local skin infection at the site of injection.
  * Ozone allergy
  * Coagulation disorders.
  * Chronic opioid use.
  * Sacroiliitis associated with disk pathology.
  * Severe ankylosing spondylitis.
  * History of corticosteroid injection within last three months.
  * Uncontrolled concomitant medical condition.
  * Severe arrhythmia, hypertensive crisis and other cardiovascular diseases.
  * Pregnant women.
  * Bowel inflammatory disease.
  * Psoriasis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-06-23 (Estimated); Primary Completion 2025-03-23 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity using visual analog scale (VAS) | 2 years
  Primary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided